CLINICAL TRIAL: NCT00502463
Title: Induction by Docetaxel/Cisplatin/5-Fluorouracil (TCF) Prior to Radiotherapy With Concomintant Cetuximab in Locally Advanced Inoperable Head and Neck Tumours - a Methodical Trial
Brief Title: Induction Chemotherapy Prior to Radio-immunotherapy in Head and Neck Cancer Stage III/IV - a Methodical Trial
Acronym: ASOG-HNO1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Austrian South Oncology Group (Network)
Collaborators: Change of sponsor 2008: new sponsor AGMT (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGMT_HNO
Record Dates: First submitted 2007-07-15; First posted 2007-07-17 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer, stage III/IV; no prior radiotherapy of head and neck region
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Docetaxel; Cisplatin; Fluorouracil; Radiotherapy; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): 3 cycles of induction chemotherapy consisting of docetaxel, cisplatin, and 5-FU followed by radiotherapy plus cetuximab
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Drug: 5-FU; Radiation: Radiotherapy; Drug: Cetuximab

INTERVENTIONS:
Drug: Docetaxel — 75mg/m² day 1
Drug: Cisplatin — 75mg/m² day 1
Drug: 5-FU — 750mg/m²/day day 1-5
Radiation: Radiotherapy — standard fraction up to a total dose of 70Gy/35 fractions/7weeks or accelerated regimen, up to a total dose of 72Gy/42 fractions over 6 weeks
Drug: Cetuximab — 250mg/m²/week after an initial loading dose of 400mg/m²

SUMMARY:
The purpose of the trial is to determine the feasibility of an induction chemotherapy with radio-immunotherapy in patients with head and neck cancer stage III/IV

DETAILED DESCRIPTION:
3 Cycles of: Docetaxel 75 mg/m2 on d1, Cisplatin 75 mg/m2 on d1, 5-FU 750 mg/m2 on days 1-5 as continuous i.v. infusion, Duration of 1 cycle: 21 days;

Followed by Cetuximab 400 mg/m2, Start of radiotherapy: 1 week after the first application of Cetuximab, During radiotherapy (35 x 2 Gy): Cetuximab 250 mg/m2 weekly, Up to 8 applications of Cetuximab.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed, locally advanced head and neck cancer
* stage III/IV
* performance status: ECOG 0-1

Exclusion Criteria:

* distant metastases
* prior radiotherapy of the head and neck region
* myocardial infarct in the last six months
* florid peptic ulcer
* neuropathy grade III/IV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-10-03 (Actual); Primary Completion 2010-01-19 (Actual); Study Completion 2014-01-19 (Actual)

PRIMARY OUTCOMES:
Locoregional tumour control | 12 months
  Time without progression of locoregional disease, locoregional recurrence of disease or death from any cause after one year.

SECONDARY OUTCOMES:
Response rate | 24 months
  PET-CT or CT, RECIST criteria
Progression free survival | 24 months
  PFS is calculated from start of therapy until disease progression or death from any cause.
Overall survival | 24 months
  OS is calculated from start of therapy to death from any cause.
Toxicities | 24 months
  The highest grade of a toxicity per patient is included in the analysis

CONTACTS AND LOCATIONS:
Overall Officials: Felix Keil, MD, Study Chair — LKH Leoben, Dept. for Hemato-Oncology
Locations (5):
- Austria (5):
  - LKH Feldkirch, Dept. of Radiooncology, Feldkirch
  - Medical University of Graz, Dept. of Radiooncology, Graz
  - LKH Leoben Dept. of Hemato-Oncology, Leoben
  - UK Salzburg, LKH: Universitätsklinik für Innere Medizin III, Salzburg
  - Medical University of Vienna, Dept. of Medicine I, Vienna

REFERENCES:
- [Result] Keil F, Selzer E, Berghold A, Reinisch S, Kapp KS, De Vries A, Greil R, Bachtiary B, Tinchon C, Anderhuber W, Burian M, Kasparek AK, Elsasser W, Kainz H, Riedl R, Kopp M, Kornek G. Induction chemotherapy with docetaxel, cisplatin and 5-fluorouracil followed by radiotherapy with cetuximab for locally advanced squamous cell carcinoma of the head and neck. Eur J Cancer. 2013 Jan;49(2):352-9. doi: 10.1016/j.ejca.2012.08.004. Epub 2012 Sep 14. PMID 22981499